CLINICAL TRIAL: NCT07126964
Title: Extended Prone Positioning for Intubated ARDS: a Randomized Controlled Trial
Brief Title: Extended Prone Positioning for Intubated ARDS
Acronym: PROSECO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: APHP240934; 2025-A00785-44 (Other: IDRCB)
Record Dates: First submitted 2025-07-29; First posted 2025-08-17 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-10

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 40-hour prone session (intervention) (Experimental): Patients will undergo PP sessions lasting for 16 hours. Maintaining PP for up to an extra 8 hours will be permitted, allowing PP sessions in the comparator group, to last a maximum of 24 hours.
  Interventions: Other: 40-hour prone session (intervention)
- 16-hour prone session (control) (Active Comparator): Patients will undergo PP sessions lasting for 16 hours. Maintaining PP for up to an extra 8 hours will be permitted, allowing PP sessions in the comparator group, to last a maximum of 24 hours.
  Interventions: Other: 16-hour prone session (control)

INTERVENTIONS:
Other: 40-hour prone session (intervention) — Patients will undergo PP sessions lasting for 16 hours. Maintaining PP for up to an extra 8 hours will be permitted, allowing PP sessions in the comparator group, to last a maximum of 24 hours.
  Arms: 40-hour prone session (intervention)
Other: 16-hour prone session (control) — Patients will undergo PP sessions lasting for 16 hours. Maintaining PP for up to an extra 8 hours will be permitted, allowing PP sessions in the comparator group, to last a maximum of 24 hours.
  Arms: 16-hour prone session (control)

SUMMARY:
Acute respiratory distress syndrome (ARDS) is an acutely induced respiratory failure characterised by the appearance of bilateral alveolar opacities on imaging and hypoxemia(1). Among strategies that have proved beneficial in terms of patient outcome, prone position (PP) is one associated with the greatest impact in terms of reduction in mortality, with PP sessions of 17h on average(2). The benefit of PP is to better homogenize the stress and strain applied to the lung by invasive ventilation. In a multicentric retrospective study involving COVID-19-related intubated ARDS patients, a strategy of extended PP, where PP was maintained for a median duration of 40 hours (h), was associated with increased survival compared to standard PP where each session lasted less than 24h(10). The main objective of this study is to investigate whether extended PP, defined as 40-hour PP sessions, can significantly reduce mortality of patients with invasively ventilated, severe ARDS, at day 28 after inclusion, compared to standard, 16-hour, PP sessions. The primary endpoint is all-cause mortality 28 days after inclusion. The study is a prospective, randomised, open-label, two-group parallel, multicenter trial comparing 40-hour extended PP to 16-hour standard PP in patients with moderate to severe ARDS. After inclusion, patients will be randomised either to standard PP, or extended PP. In the control arm, patients will be turned prone for 16-hour sessions. In the intervention arm, patients will be turned prone for 40h. In both groups, maintaining PP for up to an extra 8 hours will be permitted, allowing PP sessions to last 24 hours in the comparator group, and 48 hours in the intervention group. Inclusion criteria will be: severe ARDS, with ARDS defined according to the 2012 Berlin definition; and the severity defined as a PaO2/FiO2 ratio of <150 mm Hg, with an FiO2 of ≥ 60% persisting for at least 4h after optimization of ventilatory setting. Exclusion criteria will be : PP during the same Intensive care unit ( ICU ) stay and before inclusion, ECMO before PP, arterio-venous ECMO, persistent PaO₂/FiO₂ ratios <150 mm Hg, with FiO2 ≥ 60% on all arterial blood gases collected over a 24-hour period without prompting study inclusion, spine instability, intracranial pressure > 20 mmHg, severe brain injury, hemodynamic instability deemed to contraindicate PP by the physician in charge.

DETAILED DESCRIPTION:
Scientific justification Acute respiratory distress syndrome (ARDS) is an acutely induced respiratory failure characterised by the appearance of bilateral alveolar opacities on imaging and hypoxemia. Among strategies that have proved beneficial in terms of patient outcome, prone position (PP) is one associated with the greatest impact in terms of reduction in mortality, with PP sessions of 17h on average. The benefit of PP is to better homogenize the stress and strain applied to the lung by invasive ventilation. In a multicentric retrospective study involving COVID-19-related intubated ARDS patients, a strategy of extended PP, where PP was maintained for a median duration of 40 hours (h), was associated with increased survival compared to standard PP where each session lasted less than 24h. Our hypothesis to explain the improved survival observed with extended PP is grounded in the concept of a dose-response relationship. Maintaining patients prone beyond 24h probably augments the cumulative exposure to its beneficial effects during the initial stages of moderate to severe ARDS. This increased exposure potentially facilitates a more uniform distribution of stress and strain on the lungs during invasive ventilation, thus mitigating the risk of ventilator-induced lung injury. Additionally, we postulate that maneuvers to transition patients back to the supine position may be detrimental, potentially inducing derecruitment and exacerbating overdistension in remaining ventilated pulmonary regions. Finally, following 16-hour PP, the non-uniform distribution of strain probably immediately resumes upon patients returned in the supine position.

Design of the study The study is a prospective, randomised, open-label, two-group parallel, multicenter trial comparing 40-hour extended PP to 16-hour standard PP in patients with moderate to severe ARDS. After inclusion, patients will be randomised either to standard PP, or extended PP. In the control arm, patients will be turned prone for 16-hour sessions. In the intervention arm, patients will be turned prone for 40h. Maintaining PP for up to an extra 8-hour, will be allowed in both groups so that patients can be returned to the supine position when it is most convenient for the healthcare teams. In both groups, after randomization, positive end expiratory pressure (PEEP) will be set according to the low values of the PEEP- FiO2 table. Once back on the supine position, patients will be evaluated 6h (+/-2h) after the return on supine position (SP), or sooner in case of significant oxygenation degradation. In the absence of PP criteria, patients will be assessed: twice daily if FiO2 ≥ 60%, every time they present a significant worsening of oxygenation, and once daily if FiO2 < 60%. PP will be resume if, at any time, up to day 28, PP criteria are met, i.e. PaO2/FiO2 ratio of <150 mm Hg and PEEP set according to the PEEP-FiO2 table. The PaO2/FiO2 ratio will be analysed at the current FiO2 of the patient, not at FiO2 = 100% with an SpO2 objective between 92 and 96%.

Patients requiring inhaled NO will be kept in the protocol. Patients requiring ECMO will continue PP sessions according to their randomization arm for an extra 48 hours, corresponding to 2 standard PP sessions and one extended PP session. Afterward, subsequent PP sessions will be at the discretion of the attending physician.

For all patients, once FiO2 is < 50% a daily screening will be done to assess whether patients can be weaned from the ventilator.

Population of study participants : All patients admitted to the ICUs and intubated will be screened. We will include in the study, all patients who meet the following criteria: severe ARDS, with ARDS defined according to the 2012 Berlin definition; and the severity defined as a PaO2/FiO2 ratio of <150 mm Hg, with an FiO2 of ≥ 60% persisting for at least 4h after optimization of ventilatory setting. Optimization of ventilation setting will be done setting PEEP level to 10 cm of H2O and by optimising the level of sedation and neuromuscular blocking to obtain a volume tidal (VT) around 6 mL/kg PWB. In case of SpO2 < 92% in FiO2 = 100% and after optimization of ventilatory settings, no stabilisation period will be required before inclusion, finally, patients with persistent PaO₂/FiO₂ ratios <150 mm Hg on all arterial blood gases collected over a 24-hour period without this leading to inclusion, or inadequate protective ventilation criteria will be excluded.

Interventions or product under investigation :

Patients will undergo PP sessions lasting for 40 hours. Maintaining PP for up to an extra 8 hours will be permitted, allowing PP sessions in the intervention group, to last a maximum of 48 hours.

Comparator arm : Patients will undergo PP sessions lasting for 16 hours. Maintaining PP for up to an extra 8 hours will be permitted, allowing PP sessions in the comparator group, to last a maximum of 24 hours.

Other interventions added by the study : A one-year follow up visit will be added

Expected benefits for the participants :

The main benefit expected of extended PP is an increase in survival. As PP is a protective ventilation measure, we expect extended PP to reduce ventilator-induced lung injury which might reduce the incidence of ventilatory acquired pneumoniae and the length of stay in the ICU. It might also reduce the incidence of respiratory function sequelae after ICU discharge and overall improve post-ICU quality of life.

Expected benefits for the society:

Extended PP may lead to a reduction in the frequency of patient turning maneuvers, consequently decreasing the duration during which healthcare professionals are immobilized, in particular during night shifts when only one senior intensive care physician is available for the whole hospital.

In epidemic context, turning maneuvers have represented such a toll that teams with no ICU specialized physician where created, to whom PP was delegated. As these turning maneuvers are not without risks (incidence of accidental extubations from 0.9 to 1.25%, the presence of untrained physicians associated with non-specialized paramedical staff potentially increases the risk of severe adverse effects.

Moreover, beyond France, it has been shown that differences in ICU resources were associated with differences in COVID-19 related case fatality ratios. Improving care efficiency may be crucial for upholding care quality during periods of sudden surges of ICU patients, such as during yearly epidemic flu.

Finally, reducing the number of turning over maneuvers might help increase medical adhesion to PP. In an observational study performed during the COVID Pandemic, 25% of patients with severe ARDS were not turned prone. In more than 20% of the cases, the reason for not using PP was that hypoxemia was not severe enough. As this reason directly contradicts international guidelines, we can hypothesize that physicians are unwilling to implement a treatment whose most severe hazard is endotracheal tube and catheter dislodging. Reducing the number of maneuvers might reassure clinicians and help increase adhesion to PP.

Minimal risks and burden added by the study The most common complication associated with PP is pressure injuries. As COVID-19 patients often require several PP sessions, extending PP sessions might further increase pressure injuries cumulative incidence. A retrospective study showed that extending PP to a median of 39 h resulted in a cumulative incidence of pressure injuries of grade ≥ II of 26%. This figure is in line with the cumulative incidence of 25% described in the PROSEVA study. Okin et al (CHEST 2023) found a similar result (cumulative incidence of 30%) with PP sessions of a median of 40 h. In this latter study, more than 10% of the sessions had duration greater than 75 h. Two observational retrospective studies have shown that the cumulative incidence of grade ≥ III pressure injuries associated with extended PP remained extremely low (between 0 and 2.5%). Finally, the occurrence of pressure injuries seems to be associated with the cumulated duration of PP and not with the duration of single sessions. Long-term complications are mainly plexopathy and more specifically brachial plexus palsy. In a monocentric retrospective study, the incidence of brachial plexus palsy associated with extended PP up to 39 h was lower than the one reported with classical PP duration for COVID-19 patients. This is probably due to the non-utilization of the swimmer position in the former study.

Schedule for the study : Duration of enrolment period: 24 months Maximum period between screening and enrolment: not applicable Duration of follow-up period: 14 months Total study duration: 38 months. Exclusion period for participation in other studies: 14 months, to match the duration of follow-up period.

Number of enrolments expected per site and per month : 1,01 patient / center / month Statistical analysis : The main analysis will be in Intention to Treat (ITT) and will compare for the total population all-cause mortality between the two randomization groups. The delay for patients' survival (until day 28 after inclusion) will be analysed using a Cox proportional hazards model evaluating time to event. The event will correspond to all-cause death. Patients will be censored at the date of last news or at the end of the observation, which is 28 days after inclusion. Lost to follow-up patients will be censored at their date of last news. Covariables commonly analysed will be selected for the multivariable analysis: use of vasopressors, shock, renal replacement therapy and early use of glucocorticoids.

A Kaplan-Meier curve will be presented, stratified on the randomization group, with the 95% confidence interval (CI) of the curves. Hazard ratios will be presented with their 95% CI and tested if they are significantly different to 1. There will be no interim analysis.

ELIGIBILITY:
Inclusion Criteria:

Age of 18 years

* Admitted to ICU.
* Under invasive ventilation for a maximum of 5 days.
* Meeting the 2012 Berlin criteria for ARDS
* Protective ventilation at time of inclusion :

  1. Plateau pressure < 35 cm of H2O at the time of screening
  2. VT ≤ 8 ml/kg PBW on all nurse's charts before inclusion
  3. PEEP ≥ 5 cm H2O on all nurse's charts before inclusion

  c. Twice daily blood gas while FiO2 ≥ 60% before inclusion
* PaO2/FiO2 ≤ 150 mmHg with FiO2 ≥ 60% and Spo2 between 92 and 96% after optimization by setting PEEP to 10 mmHg, sedation levels optimization and, if necessary, administration of neuromuscular blockers to ensure patient-ventilator synchrony, with VT ≤ 8 ml/kg PBW and Pplateau < 30 cm H2O.

Exclusion Criteria:

* PP during the same ICU stay and before inclusion, ECMO before PP, arterio-venous ECMO
* persistent PaO₂/FiO₂ ratios <150 mm Hg, with FiO2 ≥ 60% on all arterial blood gases collected over a 24-hour period without this prompting study inclusion
* Spine instability, intracranial pressure > 20 mmHg, severe brain injury, hemodynamic instability deemed to contraindicate PP by the physician in charge
* Home oxygen supplementation
* Care limited to comfort measures only
* Inclusion in another interventional study including mechanically ventilated patients, which intervention concerns PP and for which mortality à D28 or D30 is the main outcome studied.
* Already included in PROSECO
* Pregnancy, subject deprived of freedom, Person under conservartorship, no insurance
* Refusal to participate expressed by the patient or his/her healthcare proxy or a close relative if present

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2025-10-18 (Actual); Primary Completion 2027-10-18 (Estimated); Study Completion 2028-10-18 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality 28 days after inclusion | 28 days after inclusion

SECONDARY OUTCOMES:
All-cause mortality 90 days after inclusion | 90 days after inclusion
The biologically confirmed ventilator associated pneumonia incidence per-1000 days of invasive ventilation | Up to day 28
Use of inhaled NO during ICU stay | Up to day 28
Use of ECMO, during ICU stay | Up to day 28
Number of days alive free of invasive ventilation at days 28 and 90 | Up to 90 days after inclusion
Number of days between inclusion and discharge from the ICU | Up to day 28
Number of days between inclusion and discharge from the hospital | Up to hospital discharge
Number of PP sessions per ICU stay (from inclusion) | Up to day 28
Total PP duration over the whole ICU stay (from inclusion), in hours | Up to day 28
28-day cost per life-years gained | Between inclusion and 28 days after inclusion
28-day cost per life saved | Between inclusion and 28 days after inclusion
90-day cost per additional ventilator-free day | Between inclusion and 90 days after inclusion
365-day cost per additional quality adjusted life year (QALY) | Between inclusion 365 days after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Thaïs Walter, Dr, Principal Investigator — University Hospital Saint-Louis Lariboisière, APHP
Locations (1):
- Hôpital Saint-Louis, Paris, France